CLINICAL TRIAL: NCT00982800
Title: Does Postoperative Gabapentin Reduce Pain, Opioid Consumption & Anxiety & Have a Positive Effect on Health Related Quality of Life After Radical Prostatectomy?
Brief Title: Does Postoperative Gabapentin Reduce Pain, Opioid Consumption and Anxiety and Have a Positive Effect on Health Related Quality of Life After Radical Prostatectomy?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Jason Sawyer, Sunnybrook Health Sciences Corporation
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 075-2005
Record Dates: First submitted 2009-09-22; First posted 2009-09-23 (Estimated); Last update posted 2010-08-06 (Estimated); Status verified 2010-08

CONDITIONS: Prostate Cancer
Keywords: gabapentin; opioid consumption; analgesic; anxiety; quality of life
MeSH Terms: conditions — Prostatic Neoplasms; Anxiety Disorders | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo Sugar Pill (Placebo Comparator): Patients are stratified based on their initial pain score in the recovery room. patients with a pain numeric rating scale of greater than or equal to 7/10 are stratified to the "high" group. then randomized to receive gabapentin 200 mg tid x 9 doses, or placebo x 9 doses. Patients with a pain score equal to or less than 6/10 are stratified to the "low" group, then randomized to receive gabapentin 200mg tid x 9 doses or placebo x 9 doses.
  All patients receive Acetaminophen 1gm every 6 hours for 3 days, Celecoxib 400mg as a loading dose then 200mg twice a day for 3 days. Patients also receive patient controlled analgesia (PCA) of hydromorphone for 24 hrs, then are transitioned to oxycodone 5-15 mg every 2 hours as needed.
  Interventions: Drug: Placebo Sugar Pill
- Gabapentin 200 mg tid x 9 doses (Active Comparator)
  Interventions: Drug: Gabapentin

INTERVENTIONS:
Drug: Gabapentin — 200mg 3x/day for 3 days (9 doses total)
  Other Names: Neurontin
  Arms: Gabapentin 200 mg tid x 9 doses
Drug: Placebo Sugar Pill
  Arms: Placebo Sugar Pill

SUMMARY:
The Acute Pain Service (APS) at Sunnybrook has been using Gabapentin 200 mg three times a day (TID) resulting in anecdotal benefits in terms of analgesia and opioid sparing effects. Higher doses of Gabapentin were associated with an increased incidence of sedation. The purpose of the study is to investigate if Gabapentin 200 mg given three times a day for 72 hours (9doses) results in a reduction in the total amount of opioid required after radical prostatectomy surgery as compared to placebo, and if analgesia is improved. This study will also examine the possible anxiety sparing effects and any health related quality of life (HRQL) changes, which may be a result of our perioperative use of gabapentin.

DETAILED DESCRIPTION:
Gabapentin Gabapentin is an anti-epileptic agent originally developed to treat spasticity (1), and eventually was found to be effective against chronic neuropathic pain (1,2). Gabapentin is available as an oral preparation and is primarily absorbed in the small intestine (1). Gabapentin is not metabolized in humans and is eliminated unchanged via the kidneys. It has no known drug-drug interactions, but it is reported that antacids can reduce the bioavailability of Gabapentin by about 20%, and Cimetidine can decrease the clearance of Gabapentin from the body by about 12% (1,2). Side effects of Gabapentin tend to be mild with somnolence (20%), dizziness (18%), ataxia (13%), and fatigue (11%) being the most common (1). The exact mechanism of Gabapentin in pain management is unknown, but it has demonstrated inhibition of mechanical hyperalgesia, and mechanical/thermal allodynia in those with neuropathic pain (1).

Over the past 5 years, there have been 20 studies examining the effect of Gabapentin on postoperative pain (1 & 3-22). All but one of these studies (16) has found that Gabapentin demonstrated a significant reduction in the amount of postoperative opioid required (16-67%) and a simultaneous reduction in pain scores. There was no difference in side effect profile between the Gabapentin and the control groups in 11 studies(3-5,7,8,10,14-16,18,20), while one(18) found a higher incidence of nausea and urinary retention in the control groups, and two studies(11,13) found a higher incidence of nausea/vomiting in the Gabapentin group. The most common side effect of increased sedation was found in only 4 studies when doses greater than 900 mg per day were given (9,11-13). The daily dose of postoperative Gabapentin in the current protocol is 200 mg TID (600 mg/day) which we currently use in our clinical population with minimal side effect issues.

There have been 8 studies looking at the administration of Gabapentin in the postoperative period (4,6-8,11,20,22,23). Fassoulaki and colleagues (6) examined pain scores and opioid consumption in postoperative breast cancer patients. Seventy-five patients undergoing surgery for breast cancer were randomized to receive Mexiletine 600 mg/day, Gabapentin 1200 mg/day or placebo for 10 days. Opioid consumption was reduced by 50% in the Gabapentin and Mexiletine groups vs. the placebo group on days 2-10. Only the Gabapentin group had decreased pain after movement from the 2nd to the 5th postoperative day. There were no adverse effects reported in the Gabapentin group. Dierking and his colleagues randomized 80 patients to receive either 1200 mg of Gabapentin or placebo 1 hr preoperatively, then either Gabapentin 600 mg or placebo at hours 8, 16, and 24 postoperatively following abdominal hysterectomies(4). Opioid consumption was reduced by 32% in this study and there was no significant difference between side effects in either group. Another study looking at postoperative outcomes and Gabapentin was published by Gilron and his colleagues who randomized 110 patients to 4 study groups: (A) placebo (B) Gabapentin 600 mg TID (C) Rofecoxib 50 mg/day (D) Gabapentin 600 mg TID & Rofecoxib 50 mg/day starting 1hr preoperatively and continuing for 72 hours postoperatively (9). This study was unique because it went further than simply looking at pain scores and morphine consumption data. Gilron and his colleagues demonstrated that the Gabapentin and the Gabapentin and Rofecoxib groups also significantly decreased movement associated pain evoked by sitting and coughing post abdominal hysterectomy. Adverse events were similar in all groups except sedation, which was more frequent with Gabapentin. Consistent with previous literature, the multimodal Gabapentin/Rofecoxib combination demonstrated opioid sparing, lower pain scores, but most importantly, decreased movement associated pain, which may be a significant factor in faster rehabilitation. In our study we have chosen to use Gabapentin 200 mg TID (bioequivalence of 600 mg/day) based on our extensive clinical experience with our patient population. This appears to be the dose at which most patients do not exhibit the Gabapentin related side effects described earlier. Only four studies have prescribed Gabapentin beyond 72 hours postoperatively (6-8,11). This is an area in which further research is needed to determine whether prolonged postoperative administration and its benefits translate into earlier hospital discharge, decreased chronic pain rates and increased functional recovery even beyond the acute post surgical time period. By following patients to 4 weeks post surgery, this study will aim to answer some of the questions regarding the perioperative use of gabapentin and its possible role ameliorating functional recovery beyond the acute hospitalization period.

The Sunnybrook Health Sciences Acute Pain Service (APS) does not know if 200 mg of Gabapentin is effective at reducing morphine consumption, and improving analgesia. Much higher doses (i.e. greater than 1800 mg/day) published in the literature were initially used at Sunnybrook, but many patients (anecdotally) became too sedated. We are currently using the dose suggested in our protocol 200 mg TID without any major problems. Therefore our goal is to assess if Gabapentin 200 mg does in fact have opioid reducing and analgesic benefits in the radical prostate population. Our pilot data from 15 patients indicates these benefits might exist. Furthermore, examining the role of gabapentin in regards to perioperative anxiety and following patients beyond the acute post surgical time period and following any changes related to their functional recovery and quality of life will help to close some of the gaps in the literature regarding the perioperative usefulness of gabapentin.

Gabapentin and Anxiety

The preoperative effectiveness of Gabapentin in decreasing anxiety scores and improving early functional recovery after anterior cruciate ligament knee surgery (n=40) has recently been demonstrated(10). Premedication with Gabapentin 1200 mg improved preoperative anxiolysis, postoperative analgesia, and early knee mobilization. By including a physical measure (active and passive knee flexion), Menigaux and colleagues also demonstrated that adequate postoperative analgesia enhances mobilization of the knee joint, thus potentially improving functional recovery. This French study examined patient's preoperative anxiety levels by administering an anxiety Visual Analogue Score prior to induction of anesthesia in the operating room. Since this method of anxiety testing has not been validated, we will use four reliable and well-validated anxiety tools in our present study. These measures are all one page questionnaires that are of little burden to patients. The anxiety measures are: The Spielberger State-Trait Anxiety Inventory, The Pain Catastrophising Scale, The Pain Anxiety Symptoms Scale and a 7 Item Modified Hospital Anxiety & Depression Scale.

The State-Trait Anxiety Inventory (STAI) consists of two self-report scales, one measuring state anxiety and the other measuring trait anxiety (24). Each scale consists of 20 statements about how the respondent may feel, and they are asked to rate how strongly they agree ("very much so") or disagree ("not at all") with the item. The S-Anxiety scale evaluates how respondents feel "right now, at this moment", whereas the T-Anxiety scale evaluates how they feel "generally". This scale has been used extensively in research and clinical practice, and has been shown to be valid and reliable (24).

Catastrophising or catastrophic thinking refers to "an exaggerated negative 'mental set' brought to bear during actual or anticipated pain experience" (25). The PCS is a 13 item self-report inventory that measures catastrophic thinking in relation to pain (26). Respondents are asked to reflect on past painful experiences and to indicate the degree to which they experience each of 13 thoughts or feelings when experiencing pain. Each item is rated on a 5-point rating scale with the end points 0 = not at all and 4 = all the time. The PCS yields a total score and three subscale scores assessing rumination (i.e., excessive focus on pain sensations), magnification (i.e., exaggerating the threat value of pain sensations) and helplessness (i.e., perceiving oneself as unable to cope with pain symptoms). The PCS has been shown to have high internal consistency {coefficient alphas: total PCS = .87, rumination = .87, magnification = .66, and helplessness = .78 (26). The PCS has been shown to predict pain intensity in patients with acute postoperative pain (27) and pain related disability in chronic neuropathic pain patients even after controlling for pain severity (28).

The Pain Anxiety Symptoms Scale (PASS) is a 40-item assessment tool that measures fear and anxiety responses to pain, and the short form of the PASS is a condensed version of the full PASS with only 20 items (29). The PASS-20 is a reliable and valid scale with adequate psychometric properties.

Finally, The Hospital Anxiety and Depression Scale (HADS, 30) is a widely used scale for measuring the symptoms of anxiety and depression among medical inpatients, outpatients and in the general population (31). The HADS is a 14-item questionnaire that measures symptoms of anxiety (7 items) and depression (7 items). For each item, the patient is asked to select from among 4 possible choices (scored from 0 to 3) the one that best describes how they have been feeling over the past week. The HADS yields an anxiety (HADS-A) and a depression (HADS-D) subscale score. We have chosen to administer only the (HADS-D) component because we feel that the other anxiety measure provide enough information in regards to anxiety. In general, the psychometric properties of the HADS are excellent. It has been administered in more than 700 studies to more than 35,000 individuals. Internal consistency for the anxiety and depression subscales show Chronbach alphas of between 0.80-0.93 for the anxiety subscale and between 0.81 and 0.90 for the depression subscale (31,32). Concurrent validity of the HADS is very good as measured by correlation coefficients of between 0.62 and 0.73 for the HADS-D with various well-validated depression scales (e.g., Beck Depression Inventory, SCL-90 Depression subscale (31,32). The HADS has been demonstrated to be sensitive to changes due to disease progression and in response to therapeutic interventions (32). The 7 item modified HADS will take less than 2 minutes to fill out (33).

The burden to patients will be minimal because all of the above measures can be completed in 15-20 minutes. Patients will be asked to complete these items at baseline (prior to surgery), on the day of hospital discharge (likely POD 3) and at the 3 month follow up post surgery.

Health Related Quality of Life

Outcomes pertaining to health related quality of life (HRQOL) are gaining importance when assessing the impact that interventions have on various disease states (34). Many tools are available, however it has been recommended that both a general and disease specific HRQOL tool be used to help ensure any changes in HRQOL status are captured (34,35). Regardless of the instrument(s) chosen they should be valid & reliable, as well as sensitive and responsive to change (35, 36). Other key considerations include utilizing a tool that captures the key dimensions of HRQOL, specifically physical, psychological, & social/role functioning (35, 37). A critical component to assessing HRQOL is that, given the subjective nature of quality of life, the data should be assessed by the patient, not the health care provider (37).

In order to meet all of these criteria, this study will utilize the SF-36 Health Outcomes questionnaire (SF-36), the UCLA Prostate Cancer Index, (UCLA-PCI) and the Brief Pain Inventory (BPI).

The SF-36 is a widely used general HRQOL tool, with extensive validity and reliability and responsiveness across many populations (38, 39). The SF-36 is a 36 question survey used to describe overall health status. It has 8 subscales (physical functioning, role limitations, bodily pain, general health perception, vitality, social function, role limitation as a result of emotional problems, and general mental health). It takes 5-10 minutes to complete and can be used with persons 14 and older.

The UCLA Prostate Cancer Index (UCLA-PCI) is also a valid and reliable tool, measuring health related outcomes specific to the prostate cancer population (40). It takes about 10 minutes to complete. In a recent review of HRQL in prostate cancer studies, the SF-36 and UCLA-PCA were the most frequently used general and disease specific tools used (41)

In order to make the measurement of pain more robust, a valid and reliable tool should be used. The Numeric Rating Scale (NRS) & Brief Pain Inventory will be used. The Brief Pain Inventory (BPI) is a widely used tool that has been validated in a wide variety of clinical and research populations, including the cancer population (42) and post operative population (43). It takes about 5 minutes to complete. The BPI measures pain intensity and pain interference on work, activity, mood, enjoyment sleep, walking, and relationships. It is important to assess baseline pain when undertaking a trial to assess pain or analgesia related outcomes.

Recently published articles have examined the effect of post operative pain on HRQOL after discharge, and have found that pain contributes to lower scores on HRQOL indices (44-46), at one week and one month post discharge.

1. Rose MA, Kam PC. Gabapentin: pharmacology and its use in pain management. Anaesthesia 2002;57:451-62.
2. Dahl JB, Mathiesen O, Moiniche S. 'Protective premedication': an option with gabapentin and related drugs? A review of gabapentin and pregabalin in the treatment of post-operative pain. Acta Anaesthesiol Scand 2004;48:1130-6.
3. Al-Mujadi H, AR, Katzarov MG et al. Preemptive gabapentin reduces postoperative pain and opioid demand following thyroid surgery. Can J Anaesth 2006;53:268-73.
4. Dierking G, Duedahl TH, Rasmussen ML et al. Effects of gabapentin on postoperative morphine consumption and pain after abdominal hysterectomy: a randomized, double-blind trial. Acta Anaesthesiol Scand 2004;48:322-7.
5. Dirks J, Fredensborg BB, Christensen D et al. A randomized study of the effects of single-dose gabapentin versus placebo on postoperative pain and morphine consumption after mastectomy. Anesthesiology 2002;97:560-4.
6. Fassoulaki A, Patris K, Sarantopoulos C, Hogan Q. The analgesic effect of gabapentin and mexiletine after breast surgery for cancer. Anesth Analg 2002;95:985-91, table of contents.
7. Fassoulaki A, Stamatakis E, Petropoulos G et al. Gabapentin attenuates late but not acute pain after abdominal hysterectomy. Eur J Anaesthesiol 2006;23:136-41.
8. Fassoulaki A, Triga A, Melemeni A, Sarantopoulos C. Multimodal analgesia with gabapentin and local anesthetics prevents acute and chronic pain after breast surgery for cancer. Anesth Analg 2005;101:1427-32.
9. Gilron I, Orr E, Tu D et al. A placebo-controlled randomized clinical trial of perioperative administration of gabapentin, rofecoxib and their combination for spontaneous and movement-evoked pain after abdominal hysterectomy. Pain 2005;113:191-200.
10. Menigaux C, Adam F, Guignard B et al. Preoperative gabapentin decreases anxiety and improves early functional recovery from knee surgery. Anesth Analg 2005;100:1394-9, table of contents.
11. Mikkelsen S, Hilsted KL, Andersen PJ et al. The effect of gabapentin on post-operative pain following tonsillectomy in adults. Acta Anaesthesiol Scand 2006;50:809-15.
12. Pandey CK, Navkar DV, Giri PJ et al. Evaluation of the optimal preemptive dose of gabapentin for postoperative pain relief after lumbar diskectomy: a randomized, double-blind, placebo-controlled study. J Neurosurg Anesthesiol 2005;17:65-8.
13. Pandey CK, Priye S, Singh S et al. Preemptive use of gabapentin significantly decreases postoperative pain and rescue analgesic requirements in laparoscopic cholecystectomy. Can J Anaesth 2004;51:358-63.
14. Pandey CK, Sahay S, Gupta D et al. Preemptive gabapentin decreases postoperative pain after lumbar discoidectomy. Can J Anaesth 2004;51:986-9.
15. Pandey CK, Singhal V, Kumar M et al. Gabapentin provides effective postoperative analgesia whether administered pre-emptively or post-incision. Can J Anaesth 2005;52:827-31.
16. Radhakrishnan M, Bithal PK, Chaturvedi A. Effect of preemptive gabapentin on postoperative pain relief and morphine consumption following lumbar laminectomy and discectomy: a randomized, double-blinded, placebo-controlled study. J Neurosurg Anesthesiol 2005;17:125-8.
17. Rorarius MG, Mennander S, Suominen P et al. Gabapentin for the prevention of postoperative pain after vaginal hysterectomy. Pain 2004;110:175-81.
18. Turan A, Karamanlioglu B, Memis D et al. Analgesic effects of gabapentin after spinal surgery. Anesthesiology 2004;100:935-8.
19. Turan A, Karamanlioglu B, Memis D et al. The analgesic effects of gabapentin after total abdominal hysterectomy. Anesth Analg 2004;98:1370-3, table of contents.
20. Turan A, Kaya G, Karamanlioglu B et al. Effect of oral gabapentin on postoperative epidural analgesia. Br J Anaesth 2006;96:242-6.
21. Turan A, Memis D, Karamanlioglu B et al. The analgesic effects of gabapentin in monitored anesthesia care for ear-nose-throat surgery. Anesth Analg 2004;99:375-8, table of contents.
22. Turan A, White PF, Karamanlioglu B et al. Gabapentin: an alternative to the cyclooxygenase-2 inhibitors for perioperative pain management. Anesth Analg 2006;102:175-81.
23. Gilron I. Review article: the role of anticonvulsant drugs in postoperative pain management: a bench-to-bedside perspective. Can J Anaesth 2006;53:562-71.
24. Spielberger CD, Gorsuch RL, Lushene R et al. State-Trait Anxiety Inventory for Adults: Manual. Palo Alto: Mind Garden, 1983.
25. Sullivan MJ, Thorn B, Haythornthwaite JA et al. Theoretical perspectives on the relation between catastrophizing and pain. Clin J Pain 2001;17:52-64.
26. Sullivan MJ, Bishop SR, Pivik J. The Pain Catastrophizing Scale: Development and Validation. Psychological Assessment 1995;7:524-32.
27. Pavlin DJ, Sullivan MJ, Freund PR, Roesen K. Catastrophizing: a risk factor for postsurgical pain. Clin J Pain 2005;21:83-90.
28. Sullivan MJ, Lynch ME, Clark AJ. Dimensions of catastrophic thinking associated with pain experience and disability in patients with neuropathic pain conditions. Pain 2005;113:310-5.
29. McCracken LM, Dhingra L. A short version of the Pain Anxiety Symptoms Scale (PASS-20): Preliminary development and validity. Pain Research and Management 2002;7:45-50.
30. Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand 1983;67:361-70.
31. Bjelland I, Dahl AA, Haug TT, Neckelmann D. The validity of the Hospital Anxiety and Depression Scale. An updated literature review. J Psychosom Res 2002;52:69-77.
32. Herrmann C. International experiences with the Hospital Anxiety and Depression Scale--a review of validation data and clinical results. J Psychosom Res 1997;42:17-41.
33. Snaith RP. The Hospital Anxiety And Depression Scale. Health Qual Life Outcomes 2003;1:29.
34. Gotay CC. Assessing cancer-related quality of life across a spectrum of applications. J Natl Cancer Inst Monogr 2004:126-33.
35. Fletcher A. Quality-of-life measurements in the evaluation of treatment: proposed guidelines. Br J Clin Pharmacol 1995;39:217-22.
36. Herr HW. Quality of life in prostate cancer patients. CA Cancer J Clin 1997;47:207-17.
37. Fossa SD. Good quality of life in prostate cancer patients: how can it be obtained? Scand J Urol Nephrol Suppl 1999;203:51-2.
38. Hopman WM, Towheed T, Anastassiades T et al. Canadian normative data for the SF-36 health survey. Canadian Multicentre Osteoporosis Study Research Group. Cmaj 2000;163:265-71.
39. Lofland JH. Measuring Patients' Health-Related Quality of LIfe: Practical Considerations for Implementing an Outcomes Management Program. P & T 2002;27:209-11.
40. Litwin MS, Hays RD, Fink A et al. The UCLA Prostate Cancer Index: development, reliability, and validity of a health-related quality of life measure. Med Care 1998;36:1002-12.
41. McNaughton-Collins M, Walker-Corkery E, Barry MJ. Health-related quality of life, satisfaction, and economic outcome measures in studies of prostate cancer screening and treatment, 1990-2000. J Natl Cancer Inst Monogr 2004:78-101.
42. Cleeland CS, Ryan KM. Pain assessment: global use of the Brief Pain Inventory. Ann Acad Med Singapore 1994;23:129-38.
43. Tittle MB, McMillan SC, Hagan S. Validating the brief pain inventory for use with surgical patients with cancer. Oncol Nurs Forum 2003;30:325-30.
44. Strassels SA, mcNicol E, Wagner AK et al. Persistent Postoperative Pain, Health-Related Quality of LIfe, and Functioning 1 Month After Hospital Discharge. Acute Pain 2004;6:95-104.
45. Wu CL, Naqibuddin M, Rowlingson AJ et al. The effect of pain on health-related quality of life in the immediate postoperative period. Anesth Analg 2003;97:1078-85, table of contents.
46. VanDenKerkhof EG, Hopman WM, Towheed T et al. Pain, health-related quality of life and health care utilization after inpatient surgery: a pilot study. Pain Res Manag 2006;11:41-7.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing radical prostatectomy
* Able to read and write english (assistance is allowed)
* Normal creatinine blood serum level
* No known allergies to study medications

Exclusion Criteria:

* Patients not providing informed consent
* Patients less than 18 years of age or greater than 75 years of age
* Known allergy to any of the medications being used
* History of drug or alcohol abuse
* Preoperative pain
* Patients unable or unwilling to use PCA
* Patients with impaired renal function (Creatinine >106)

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2007-06; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Will Gabapentin 200mg TID have pain and opioid sparing effects? | 3 days after surgery

SECONDARY OUTCOMES:
Does postoperative Gabapentin have perioperative anxiety sparing effects and do these effects last beyond hospital discharge? | up to 1 month postoperatively
3. Will improved analgesia with Gabapentin facilitate recovery and demonstrate effects on health related quality of life? | up to 1 month postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Colin McCartney, MD, Study Chair — Sunnybrook Health Sciences Center
Locations (1):
- Sunnybrook Health Sciences Center, Toronto, Ontario, Canada